CLINICAL TRIAL: NCT03394833
Title: Hemodynamic Stability During an Induction of Anaesthesia: A Randomized, Non-blinded Study
Brief Title: Hemodynamic Stability During Induction of Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tomi Myrberg, Principal Investigator, Umeå University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016/361-31
Record Dates: First submitted 2017-11-17; First posted 2018-01-09 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Hemodynamic Instability; Fluid Therapy; Anesthesia; Adverse Effect
Keywords: preoperative; fluid therapy; hemodynamics; anesthesia induction; rapid sequence induction; TCI
MeSH Terms: interventions — Polygeline

STUDY DESIGN:
Intervention Model Description: Non-blinded randomization. Standardized method comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative fluids (Experimental): 40 individuals receiving preoperative colloid fluid bolus at 6 ml/kg LBW, (Gelofusine™, Fresenius Kabi AB, Sweden) before anesthesia induction by TCI (n = 20) or RSI (n =20).
  Interventions: Other: gelofusine
- No preoperative fluids (No Intervention): 40 individuals anesthetized by TCI (n = 20) or RSI (n =20) without preoperative fluids.

INTERVENTIONS:
Other: gelofusine — Preoperative colloid fluid bolus 6ml/kg ideal body weight
  Other Names: colloid fluid
  Arms: Preoperative fluids

SUMMARY:
The study aim is to investigate if preoperative volume bolus based on lean body weight could preserve mean arterial pressure during target controlled infusion of anaesthesia (TCI) or rapid sequence induction of anaesthesia (RSI) in non-cardiac, non-morbidly obese surgery.

DETAILED DESCRIPTION:
40 individuals are enrolled to TCI and RSI groups respectively. The randomization process for preoperative fluid bolus prior to induction of anaesthesia is conducted in respective group at the day of surgery. Preoperative colloid fluid therapy (6 ml/kg LBW, Gelofusine™, Fresenius Kabi Ab, Sweden) is infused rapidly before non-invasive baseline blood pressure (NIBP) measurements in twenty individuals in each group. No other intravenous fluids before induction of anaesthesia.

NIBPs, pulse frequency, peripheral saturation (SpO2) are registered and collected 20 minutes post induction.

ELIGIBILITY:
Inclusion Criteria:

* 80 individuals over 18 years, body mass index ≤ 35 kg/m2, electively scheduled for breast cancer surgery, endocrinologic surgery (thyroid, parathyroid) and general abdominal surgery.

Exclusion Criteria:

* instable angina pectoris at the day of surgery, severe bronchial asthma or COPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of blood pressure drops | 20 minutes post anesthesia induction
  blood pressure drop below mean arterial pressure at 65 mmHg during anesthesia induction
Effect of preoperative fluid bolus | 20 minutes post anesthesia induction
  Does preoperative fluid bolus decrease incidence of blood pressure drops

CONTACTS AND LOCATIONS:
Overall Officials: Tomi P Myrberg, MD PhD, Principal Investigator — Umeå University, Norrbotten county concil
Locations (1):
- Sunderby hospital, Luleå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myrberg T, Lindelof L, Hultin M. Effect of preoperative fluid therapy on hemodynamic stability during anesthesia induction, a randomized study. Acta Anaesthesiol Scand. 2019 Oct;63(9):1129-1136. doi: 10.1111/aas.13419. Epub 2019 Jun 26. PMID 31240711